CLINICAL TRIAL: NCT03730025
Title: Impact of a Mobile Application for Heart Rate Assessment in Simulated Neonatal Resuscitation: a Randomized Controlled Crossover Study
Brief Title: Impact of a Mobile Application for Heart Rate Assessment in Simulated Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Novara2
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Resuscitation; Heart Rate Assessment
Keywords: Heart rate; Assessment; Time; Resuscitation intervention
MeSH Terms: interventions — Auditory Perception

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auscultation plus NeoTapAS (Experimental): Pediatric resident responsible for HR assessment will estimate the HR by listening to the praecordium with a stethoscope. When using NeoTapAS, he/she will simultaneously tap the same pace on the screen of an iPad with the NeoTapAS app installed and will verbally communicate the HR displayed on the screen.
  Interventions: Other: Auscultation plus NeoTapAS
- Auscultation without NeoTapAS (Active Comparator): Pediatric resident responsible for HR assessment will mentally calculate the HR based on auscultation (by counting the number of beats in 6 seconds and multiplying by 10) and will verbally communicate the calculated HR.
  Interventions: Other: Auscultation without NeoTapAS

INTERVENTIONS:
Other: Auscultation plus NeoTapAS — Pediatric resident responsible for HR assessment will estimate the HR by listening to the praecordium with a stethoscope. When using NeoTapAS, he/she will simultaneously tap the same pace on the screen of an iPad with the NeoTapAS app installed and will verbally communicate the HR displayed on the screen.
  Arms: Auscultation plus NeoTapAS
Other: Auscultation without NeoTapAS — Auscultation without NeoTapAS
  Arms: Auscultation without NeoTapAS

SUMMARY:
NeoTapAdvancedSupport (NeoTapAS) is a free-of-charge mobile application that showed good accuracy in HR estimation. This study aims to evaluate the impact of NeoTapAS on timing of HR communication and of resuscitation interventions in a high fidelity simulation scenario.

DETAILED DESCRIPTION:
Assessing the HR by auscultation can be limited due to imprecise auscultation and/or errors in mental computation, leading to inappropriate or delayed resuscitation. Previous studies evaluated a free-of-charge mobile application (NeoTapAdvancedSupport, NeoTapAS) to help HR assessment in a simulated scenario of neonatal resuscitation. NeoTapAS showed good accuracy in estimating HR and could be a useful tool in resource-constrained settings.

Another potential advantage of using NeoTapAS may be the anticipation of HR communication during resuscitation, because it avoids mental computation and possible errors due to the stressful situation. In addition, prompt HR assessment may lead to anticipating resuscitation interventions. However, these hypotheses remain to be demonstrated.

The aim of this study is to evaluate the promptness in HR communication using NeoTapAS compared with mental computation in a high-fidelity simulated newborn resuscitation scenario. In addition, the impact of NeoTapAS on timing of resuscitation procedures will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric residents from third to fifth year of residency of the University of Piemonte Orientale who were trained on neonatal resuscitation

Exclusion Criteria:

* Lack of EC approval
* Lack of consent to record the scenario and to use the data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Timing of the first HR communication. | 1 min
  Time elapsed from birth to the first HR communication

SECONDARY OUTCOMES:
Timing of the second HR communication | 2 min
Timing of the third HR communication | 3 min
Timing of the fourth HR communication | 4 min
Timing of resuscitation interventions (positive pressure ventilation, chest compressions, intubation and administration of first dose of adrenaline | 10 min
Timing of the fifth HR communication | 5 min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Piemonte Orientale, Novara, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Binotti M, Cavallin F, Ingrassia PL, Pejovic NJ, Monzani A, Genoni G, Trevisanuto D. Heart rate assessment using NeoTapAdvancedSupport: a simulation study. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F440-F442. doi: 10.1136/archdischild-2018-315408. Epub 2018 Sep 27. PMID 30262463
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Background] Myrnerts Hook S, Pejovic NJ, Marrone G, Tylleskar T, Alfven T. Accurate and fast neonatal heart rate assessment with a smartphone-based application - a manikin study. Acta Paediatr. 2018 Sep;107(9):1548-1554. doi: 10.1111/apa.14350. Epub 2018 Apr 22. PMID 29604115
- [Background] Murphy MC, De Angelis L, McCarthy LK, O'Donnell CPF. Comparison of infant heart rate assessment by auscultation, ECG and oximetry in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F490-F492. doi: 10.1136/archdischild-2017-314367. Epub 2018 May 25. PMID 29802102
- [Background] Chitkara R, Rajani AK, Oehlert JW, Lee HC, Epi MS, Halamek LP. The accuracy of human senses in the detection of neonatal heart rate during standardized simulated resuscitation: implications for delivery of care, training and technology design. Resuscitation. 2013 Mar;84(3):369-72. doi: 10.1016/j.resuscitation.2012.07.035. Epub 2012 Aug 25. PMID 22925993
- [Derived] Cavallin F, Binotti M, Ingrassia PL, Genoni G, Rizzollo S, Monzani A, Trevisanuto D. Impact of a mobile application for heart rate assessment in simulated neonatal resuscitation: a randomised controlled cross-over study. Arch Dis Child Fetal Neonatal Ed. 2020 Jan;105(1):41-44. doi: 10.1136/archdischild-2018-316757. Epub 2019 May 17. PMID 31101662